CLINICAL TRIAL: NCT01519453
Title: Reducing Asthma Morbidity in High Risk Minority Preschool Children (Asthma Basic Care (ABC) at Head Start)
Brief Title: Reducing Asthma Morbidity In High Risk Minority Preschool Children
Acronym: ABC-HS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00046455; HL-107223 (Other Grant/Funding Number: National Heart, Lung, and Blood Institute)
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Asthma
Keywords: Asthma; Preschool; Health Disparities; Implementation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Based Asthma Education (Experimental): Families will receive 4 home based and 3 phone based asthma education sessions with a community asthma outreach worker
  Interventions: Behavioral: Home Based Asthma Education
- Control (No Intervention): There is no control arm specific intervention

INTERVENTIONS:
Behavioral: Home Based Asthma Education — 4 home based and 3 phone based sessions with community asthma outreach worker to provide families with asthma education
  Arms: Home Based Asthma Education

SUMMARY:
Low-income, minority children are disproportionately affected by asthma and can experience higher rates of asthma attacks, lower lung function, decreased physical activity, increases in school absenteeism, and higher rates of death. The National Center for Children in Poverty suggests that effective interventions to improve asthma and reduce harm for high risk groups (like low-income minority children) must begin in early childhood. Previous research has shown that asthma education programs can be effective to improve overall asthma management in preschool children, but there has been limited sustainability of these programs in medical, educational, and social environments that serve young high risk children. One of the core missions of federally-funded Head Start programs is to provide preventive health services and screening to their low-income preschool students and would be an ideal setting in the community to disseminate an early asthma education program. The purpose of this study is to draw on our health and research partnership with Baltimore City Head Start programs to test the effectiveness of a home-based asthma education intervention combined with a Head Start level asthma education program compared to a Head Start level asthma education program alone.

DETAILED DESCRIPTION:
Despite advances in asthma therapies and the wide-spread dissemination of asthma clinical guidelines, low-income, minority children have disproportionately high morbidity and mortality from asthma. The National Center for Children in Poverty has strongly argued that effective interventions to improve asthma health disparities and reduce harm must begin in early childhood. Previous efficacy studies have suggested that asthma education programs can be effective in improving overall management of asthma for preschool children. However, for these promising asthma intervention strategies to have sustainable public health impact for low-income, minority children they must be integrated within those medical, educational and social structures that serve these young high risk children, such as community clinics, schools and day care programs. Because one of the core missions of federally-funded Head Start programs is to provide preventive health services and screening to their low-income preschool students, Head Start represents an ideal community setting for disseminating early asthma education. The investigators propose to draw on our established health and research partnership with Head Start programs in Baltimore City to test the effectiveness of this home-based asthma education intervention with demonstrated efficacy, when delivered in the context of a Head Start-wide asthma education program. The investigators further propose to partner with Head Start to support and evaluate adoption, maintenance and dissemination of new knowledge gained from this project. Specifically the investigators hypothesize that participants receiving the ABC intervention combined with a HS-level asthma education will have more symptom free days at the 6-, 9-, and 12-month evaluation when compared with participants in the HS-level asthma education alone. The investigators plan to enroll of 406 children age 2-6 years old enrolled in Head Start with symptomatic asthma. Secondary outcome measures include other measures of asthma morbidity (i.e., hospitalizations, Emergency Department visits, oral steroid bursts, school absences, and caregiver quality of life). The investigators will also evaluate the mediating effects of outcomes expectancies, self-efficacy, asthma knowledge, motivation, and asthma management practices, as well as moderator effects, such as health literacy, caregiver depression, neighborhood cohesion, family management of asthma, and Head Start adoption and dissemination of an asthma education curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Head Start
* Physician diagnosed asthma or reactive airway disease
* Resides in Baltimore City or Baltimore County
* English Speaking

Exclusion Criteria:

* Enrolled in another pulmonary research study
* Sibling enrolled in study

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 404 (Actual)
Dates: Start 2011-09; Primary Completion 2017-11 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Rand, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual participant data with other researchers

REFERENCES:
- [Background] Callaghan-Koru JA, Riekert KA, Ruvalcaba E, Rand CS, Eakin MN. Home Medication Readiness for Preschool Children With Asthma. Pediatrics. 2018 Sep;142(3):e20180829. doi: 10.1542/peds.2018-0829. Epub 2018 Aug 7. PMID 30087197
- [Background] Ruvalcaba E, Chung SE, Rand C, Riekert KA, Eakin M. Evaluating the implementation of a multicomponent asthma education program for Head Start staff. J Asthma. 2019 Feb;56(2):218-226. doi: 10.1080/02770903.2018.1443467. Epub 2018 Mar 15. PMID 29543493
- [Background] Sadreameli SC, Riekert KA, Matsui EC, Rand CS, Eakin MN. Family Caregiver Marginalization is Associated With Decreased Primary and Subspecialty Asthma Care in Head Start Children. Acad Pediatr. 2018 Nov-Dec;18(8):905-911. doi: 10.1016/j.acap.2018.04.135. Epub 2018 May 3. PMID 29730244
- [Result] Eakin MN, Zaeh S, Eckmann T, Ruvalcaba E, Rand CS, Hilliard ME, Riekert KA. Effectiveness of a Home- and School-Based Asthma Educational Program for Head Start Children With Asthma: A Randomized Clinical Trial. JAMA Pediatr. 2020 Dec 1;174(12):1191-1198. doi: 10.1001/jamapediatrics.2020.3375. PMID 33016987
- [Derived] Lu MA, Eckmann T, Ruvalcaba E, McQuaid EL, Rand CS, Riekert KA, Eakin MN. Family management of asthma in Head Start preschool children. Ann Allergy Asthma Immunol. 2022 Feb;128(2):178-183. doi: 10.1016/j.anai.2021.11.002. Epub 2021 Nov 10. PMID 34774736

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 refused to complete a baseline assessment after consent
  1 participant dropped due to no asthma after consent
  3 families were pilot participants and their data is not represented in final outcomes except in sponsor reporting
Groups:
- Home Based Asthma Education Arm: This arm consists of caregiver and child pairs. Caregiver is consented and is asked questions relating to the child's health due to young age of child.
  For those randomly assigned to the Home Based Asthma Education Arm- the consented caregiver received 4 home based and 3 phone based asthma education sessions with a community asthma outreach worker. Due to age of child, primary asthma management is provided by the caregiver, so intervention was delivered directly to caregiver.
- Control Arm: This arm consists of caregiver and child pairs. Caregiver is consented and is asked questions relating to the child's health due to young age of child.
  Caregiver is not provided a control arm specific intervention.
Period: Overall Study
Arm/Group | Home Based Asthma Education Arm | Control Arm
Started | 199 (Number of dyads (caregiver-child pairs) or 398 individuals) | 199 (Number of dyads (caregiver-child pairs) or 398 individuals)
3 Month | 160 (Number of dyads (caregiver-child pairs) or 320 individuals) | 181 (Number of dyads (caregiver-child pairs) or 362 individuals)
6 Month | 153 (Number of dyads (caregiver-child pairs) or 306 individuals) | 175 (Number of dyads (caregiver-child pairs) or 350 individuals)
9 Month | 159 (Number of dyads (caregiver-child pairs) or 318 individuals) | 166 (Number of dyads (caregiver-child pairs) or 332 individuals)
Completed (Number completing 12 month follow up assessment) | 147 (Number of dyads (caregiver-child pairs) or 294 individuals) | 163 (Number of dyads (caregiver-child pairs) or 326 individuals)
Not Completed | 52 | 36

BASELINE CHARACTERISTICS:
Population: There were 199 caregiver-child pairs in each arm.
Groups:
- Home Based Asthma Education: This arm consists of caregiver and child pairs. Caregiver is consented and is asked questions relating to the child's health due to young age of child.
  For those randomly assigned to the Home Based Asthma Education Arm- the consented caregiver received 4 home based and 3 phone based asthma education sessions with a community asthma outreach worker. Due to age of child, primary asthma management is provided by the caregiver, so intervention was delivered directly to caregiver.
- Control: This arm consists of caregiver and child pairs. Caregiver is consented and is asked questions relating to the child's health due to young age of child.
  Caregiver is not provided a control arm specific intervention.
- Total: Total of all reporting groups
Arm/Group | Home Based Asthma Education | Control | Total
Number analyzed (Participants) | 199 | 199 | 398
Age, Categorical [Count of Participants; unit: Participants]
  Child in caregiver-child pair: <=18 years | 199 | 199 | 398
  Child in caregiver-child pair: Between 18 and 65 years | 0 | 0 | 0
  Child in caregiver-child pair: >=65 years | 0 | 0 | 0
  Caregiver in caregiver-child pair: <=18 years | 0 | 0 | 0
  Caregiver in caregiver-child pair: Between 18 and 65 years | 199 | 198 | 397
  Caregiver in caregiver-child pair: >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years]
  Child in caregiver-child pair | 4.2 (0.6) | 4.2 (0.8) | 4.2 (0.7)
  Caregiver in caregiver-child pair | 30.9 (7.8) | 31.9 (8.9) | 31.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Child in caregiver-child pair: Female | 76 | 75 | 151
  Child in caregiver-child pair: Male | 123 | 124 | 247
  Caregiver in caregiver-child pair: Female | 184 | 187 | 371
  Caregiver in caregiver-child pair: Male | 15 | 12 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Data provided here refer to child in caregiver-child pair. Ethnicity of enrolled caregiver was not collected.
  Participants
    Child in caregiver-child pair: Hispanic or Latino | 6 | 8 | 14
    Child in caregiver-child pair: Not Hispanic or Latino | 193 | 191 | 384
    Child in caregiver-child pair: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Data provided here refer to child in caregiver-child pair. Race of enrolled caregiver was not collected.
  Participants
    Child in caregiver-child pair: American Indian or Alaska Native | 0 | 0 | 0
    Child in caregiver-child pair: Asian | 0 | 0 | 0
    Child in caregiver-child pair: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Child in caregiver-child pair: Black or African American | 189 | 190 | 379
    Child in caregiver-child pair: White | 4 | 4 | 8
    Child in caregiver-child pair: More than one race | 2 | 5 | 7
    Child in caregiver-child pair: Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 199 | 199 | 398

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control as Determined by Test for Respiratory and Asthma Control in Kids Assessment Tool
Description: The Test for Respiratory and Asthma Control in Kids test is an assessment tool consisting of 5 questions posed to caregivers and designed to assess respiratory and asthma control in patients between 12 months and 5 years. It addresses risk and impairment domains outlined in the Asthma Guidelines and is meant to be interpreted by medical professionals. A total score is calculated from 0-100 with scores less than 80 indicating the child's asthma may not be under control and scores of 80 or more indicating that a child's asthma seems to be under control.
Time Frame: Baseline, 3, 6, 9 and 12 months
Population: Participants analyzed represent children with asthma enrolled in the protocol as caregiver-child pairs. Number analyzed per row vary since some families were unable to be contacted for specific assessment time points, but were able to be contacted for future assessments.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Home Based Asthma Education | Control
Number analyzed (Participants) | 199 | 199
score on a scale
  Baseline | 70 [50 to 80] | 75 [55 to 85]
  3 months: number analyzed (Participants) | 160 | 181
  3 months | 85 [70 to 95] | 80 [60 to 90]
  6 months: number analyzed (Participants) | 153 | 175
  6 months | 85 [75 to 95] | 85 [70 to 95]
  9 months: number analyzed (Participants) | 159 | 166
  9 months | 85 [65 to 95] | 85 [75 to 95]
  12 months: number analyzed (Participants) | 147 | 163
  12 months | 85 [70 to 95] | 85 [75 to 95]

2. Secondary Outcome: Total Number of Emergency Department (ED) Visits [Child]
Description: Aggregate number of ED visits for asthma in past 90 days for all participants.
Time Frame: Baseline, 3, 6, 9 and 12 months
Population: as for outcome 1
Measure: Number; unit: ED visits
Arm/Group | Home Based Asthma Education | Control
Number analyzed (Participants) | 199 | 199
ED visits
  Baseline | 65 | 50
  3 months: number analyzed (Participants) | 160 | 181
  3 months | 34 | 42
  6 months: number analyzed (Participants) | 153 | 175
  6 months | 28 | 32
  9 months: number analyzed (Participants) | 159 | 166
  9 months | 37 | 38
  12 months: number analyzed (Participants) | 147 | 163
  12 months | 31 | 35

3. Secondary Outcome: Total Number of Hospitalizations [Child]
Description: Aggregate number of hospitalizations due to asthma 12 months before randomization vs after randomization for all participants.
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Number; unit: asthma related hospitalizations
Arm/Group | Home Based Asthma Education | Control
Number analyzed (Participants) | 199 | 199
asthma related hospitalizations
  Baseline | 6 | 10
  12 months: number analyzed (Participants) | 147 | 163
  12 months | 7 | 24

ADVERSE EVENTS:
Time Frame: 12 months.
Description: Reportable Adverse Events included: Deaths of child or consented caregiver, Asthma related hospitalization for child or consented caregiver, formal complaint about study, any psychosocial adverse event related to the study intervention, or any other potential adverse event as identified by Principal Investigator.
  Note: 199 child/consented caregiver pairs were enrolled making a total of 398 per arm assessed for adverse events.
Arm/Group | Home Based Asthma Education | Control
All-Cause Mortality (participants affected / at risk) | 0/398 | 0/398
Serious Adverse Events (participants affected / at risk) | 8/398 | 16/398
Other Adverse Events (participants affected / at risk) | 2/398 | 0/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Home Based Asthma Education (N=398) | Control (N=398)
Hospitalization due to asthma [child] (Respiratory, thoracic and mediastinal disorders) | 6/199 (9) | 14/199 (24)
Non asthma related hospitalization [child] (Blood and lymphatic system disorders) | 0/199 (0) | 1/199 (1)
Hospitalization due to asthma [consented caregiver] (Respiratory, thoracic and mediastinal disorders) | 2/199 (2) | 2/199 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Home Based Asthma Education (N=398) | Control (N=398)
Psychosocial Event [consented caregiver] (Social circumstances) | 2/199 (2) | 0/199 (0) — Psychosocial events included call to child protective services due to young child left home unattended and a consented caregiver becoming very emotional and upset during survey due to past events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT01519453/Prot_SAP_000.pdf